CLINICAL TRIAL: NCT02437409
Title: Acute Recanalization of Thrombo-Embolic Ischemic Stroke With pREset (ARTESp)
Acronym: ARTESp
Status: Completed | Type: Observational
Sponsor: Phenox GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: T01-072012
Record Dates: First submitted 2015-04-28; First posted 2015-05-07 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-07

CONDITIONS: Stroke
Keywords: Ischemic, Acute
MeSH Terms: conditions — Stroke; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: pREset thrombectomy retriever — Interventional recanalization of acute cerebral vessel occlusions with the pREset thrombectomy system alone or in combination with intravenous or intraarterial thrombolytics (rt-PA).

SUMMARY:
ARTESp is a prospective multicenter study in which the pREset thrombectomy system (phenox GmbH* Germany) will be examined. The effectiveness, safety and the long-term success when using the pREset to treat acute occlusions of cerebral vessels will be analyzed.

*German: "Gesellschaft mit beschränkter Haftung", limited liability company

DETAILED DESCRIPTION:
ARTESp is a prospective multicenter study in which the pREset thrombectomy system (phenox GmbH Germany) will be examined. The effectiveness, safety and the long-term success when using the pREset to treat acute occlusions of cerebral vessels will be analyzed.

In this study the market-approved, self-expandable stent retriever (pREset, phenox GmbH, Germany) will be used to achieve a direct flow recovery.

The thrombectomy system will be unfolded directly in the vessel occlusion. In a second step, the system and the thrombus will be pulled back into the guide catheter.

It is planned to enroll 100 patients at the age of 18 until 85 years, with a NIHSS (National Institutes of Health Stroke Scale) ≥ 8 and ≤ 30. The preconditions for study enrollment are the written consent of the patient or of the legal representative and the fulfillment of all mentioned inclusion and exclusion criteria. Pregnant women are excluded from study participation.The clinical interventions are in accordance with the clinical standard of care for the treatment of this patient population.

The mRS (Modified Rankin Scale) on day 30, the NIHSS on day 90 and an imaging procedure on day 90 may be performed by the study site provided that it corresponds to the clinical standards of the study site.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 and ≤ 85 years.
* Patients with acute-onset stroke in the 0-6 hour time window for cerebral onset of symptoms and in angiography with a TICI reperfusion (Thrombolysis in Cerebral Infarction) value of 0 or 1 of at least one major cerebral artery (carotid artery, A. media , anterior cerebral artery, basilar artery, vertebral artery, posterior cerebral artery).
* NIHSS (National Institutes of Health Stroke Scale) ≥ 8
* Signed Informed Consent by patient / legal representative to participate in the study.

Exclusion Criteria:

* Pregnancy
* Demarcated infarcted area in the initial Cranial CT or intracranial haemorrhage,
* Rapid improvement of neurological symptoms
* NIHSS > 30
* Anticoagulation with warfarin with INR (international normalized ratio) > 3.0,
* Platelets <30,000,
* Glucose <50mg/dl,
* Life expectancy <90 days

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients harboring an acute ischemic stroke in at least one of the major intracranial arteries
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Reith, Prof., Principal Investigator — Universitätsklinikum des Saarlands
Locations (4):
- Germany (4):
  - Katharinenhospital, Stuttgart, Baden-Wurttemberg
  - Klinikum rechts der Isar, München, Bavaria
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsklinikum des Saarlandes, Homburg, Saarland

REFERENCES:
- [Derived] Prothmann S, Schwaiger BJ, Gersing AS, Reith W, Niederstadt T, Felber A, Kurre W. Acute Recanalization of Thrombo-Embolic Ischemic Stroke with pREset (ARTESp): the impact of occlusion time on clinical outcome of directly admitted and transferred patients. J Neurointerv Surg. 2017 Sep;9(9):817-822. doi: 10.1136/neurintsurg-2016-012556. Epub 2016 Aug 16. PMID 27530601
- See also: phenox GmbH — http://www.phenox.info

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 115 patients started the study, but little by little, 15 patients were excluded/discontinued due to screening failure or withdrawn consent.
Pre-assignment Details: No assignment to groups was performed due to single-arm study.
Groups:
- All Patients: Treated with pREset Thrombectomy Retriever
Period: Overall Study
Arm/Group | All Patients
Started | 115 (Eventually 100 evaluable patients, attrition rate of 15%)
Completed | 100 (In total 100 patients fulfilled the in-and exclusion criteria,15 patients were excluded/discontinued)
Not Completed | 15
Not completed — Withdrawal by Subject | 3
Not completed — Screening failure | 12

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender
  Participants
    Female | 55
    Male | 45
Region of Enrollment [Number; unit: participants]
  Germany | 100

OUTCOME MEASURES:

1. Primary Outcome: Neurological Condition of the Patient
Description: modified Rankin Scale (mRS)
  Neurological Condition is measured by the "Modified Rankin Scale (mRS)". This scale ranges from 0 - 6:
  0 = No symptoms at all;
  1. = able to carry out all usual duties and activities;
  2. = unable to carry out all previous activities, but able to look after own affairs without assistance;
  3. = requiring some help, but able to walk without assistance;
  4. = unable to walk without assistance and unable to attend to own bodily needs without assistance;
  5. = bedridden, incontinent and requiring constant nursing care and attention;
  6. = dead
Time Frame: 90 days after treatment
Population: All Patients
Measure: Number; unit: patients
Arm/Group | All Patients
Number analyzed (Participants) | 100
patients
  mRS 0 | 23
  mRS 0-1 | 52
  mRS 0-2 | 60
  mRS 3-5 | 29
  mRS 6 | 7
  Lost to follow-up | 4

2. Secondary Outcome: Neurological Condition of the Patient
Description: The National Institutes of Health Stroke Scale (NIHSS) is a commonly used measure to assess the severity of a stroke. All items are rated and scores are added at the end. A higher score corresponds to a more severe stroke. Assessed are:
  1. Level of Conciousness (LOC) (0-3) 1a. LOC Questions (0-2) 1b. LOC Commands (0-2)
  2. Best Gaze (0-2)
  3. Visual (0-3)
  4. Facial palsy (0-3)
  5. Motor arm (0-4)
  6. Motor leg (0-4)
  7. Limb ataxia (0-2)
  8. Sensory (0-2)
  9. Best Language (0-3)
  10. Dysarthria (0-2)
  11. Extinction and Inattention (0-2)
  CLASSIFICATION:
  0 No stroke symptoms 1-4 Minor stroke 5-15 Moderate stroke 16-20 Moderate to severe stroke 21-42 Severe stroke
  As published by ninds.nih.gov: http://www.ninds.nih.gov/doctors/NIH_Stroke_Scale.pdf
Time Frame: 24 to 72 hr after treatment
Population: All Patients
Measure: Median (Full Range); unit: NIHSS score
Arm/Group | All Patients
Number analyzed (Participants) | 100
NIHSS score | 5 [0 to 42]

3. Secondary Outcome: Intracranial Hemorrhage (ICH)
Description: Intracranial hemorrhage was assessed via imaging material (e.g. Digital Subtraction Angiography - DSA or CT) as forwarded by the clinical sites.
Time Frame: 24 hr after treatment
Population: All Patients
Measure: Number; unit: patients
Arm/Group | All Patients
Number analyzed (Participants) | 100
patients | 14

4. Secondary Outcome: Time From Groin Puncture to Recanalization
Time Frame: during intervention, up to 3 hr
Population: All Patients
Measure: Median (Full Range); unit: minutes
Arm/Group | All Patients
Number analyzed (Participants) | 100
minutes | 40 [6 to 159]

5. Secondary Outcome: Recanalization of the Target Vessel
Description: original Thrombolysis in Cerebral Infarction score (o-TICI) The TICI scale indicates perfusion of an occluded blood vessel, it is used in angiographic imaging.
  Grade 0 = no perfusion Grade 1 = Penetration with minimal perfusion. The contrast material passes beyond the area of obstruction but fails to opacify the entire cerebral bed distal to the obstruction for the duration of the angiographic run, Grade 2a = Only partial filling (<2/3) of the entire vascular territory is visualized, Grade 2b = Complete filling of all of the expected vascular territory is visualized, but the filling is slower than normal, Grade 3 = complete perfusion.
Time Frame: at the end of intervention, up to 3 hr
Population: 100 patients harboured 109 vessel occlusions
Measure: Number; unit: number of vessels
Units Other Than Participants: vessel occlusions
Groups:
- Occluded Vessels: 100 patients harboured 109 vessel occlusions
Arm/Group | Occluded Vessels
Number analyzed (Participants) | 100
Number analyzed (vessel occlusions) | 109
number of vessels
  TICI 0 | 7
  TICI 1 | 2
  TICI 2a | 8
  TICI 2b | 40
  TICI 3 | 52

6. Secondary Outcome: No. of Passages Needed to Reach the Final TICI Score With pREset
Time Frame: during intervention, up to 3 hr
Population: 100 patients harboured 109 vessel occlusions
Measure: Mean (Standard Deviation); unit: passes
Units Other Than Participants: vessel occlusions
Arm/Group | Occluded Vessels
Number analyzed (Participants) | 100
Number analyzed (vessel occlusions) | 109
passes | 1.7 (0.96)

ADVERSE EVENTS:
Time Frame: 90 days after procedure
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 7/100
Other Adverse Events (participants affected / at risk) | 24/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=100)
Mortality (Injury, poisoning and procedural complications) | 7 (7) — Led to death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=100)
Extravasation (Vascular disorders) | 2 (2)
Vasospasm (Vascular disorders) | 3 (3)
Emboli to a new territory (Vascular disorders) | 2 (2)
Emboli to the same territory (Vascular disorders) | 3 (3)
Focal subarachnoid hemorrhages around the target vessel (Vascular disorders) | 7 (7)
PH I (Vascular disorders) | 4 (4)
PH II (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data must only be published after completion of the study. Publication of e.g. single center experience within the study is not allowed until the aggregate data have been submitted.

All information and data generated in association with this study will be held in strict confidence and remain in the sole property of phenox GmbH. The investigator agrees to use this information for the sole purpose of completing this study and for no other purpose without written consent from phenox GmbH.